CLINICAL TRIAL: NCT01277081
Title: To Assess the Subjective Effect of Two Paracetamol Preparations on the Feeling of Breathing in Subjects With the Common Cold.
Brief Title: Effect of Paracetamol on the Common Cold
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C7100991
Record Dates: First submitted 2011-01-12; First posted 2011-01-14 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2013-06

CONDITIONS: Common Cold
Keywords: Paracetamol; Common cold
MeSH Terms: conditions — Common Cold | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol hot drink (Active Comparator): Hot drink containing paracetamol
  Interventions: Drug: Paracetamol hot drink
- Paracetamol tablets (Active Comparator): Paracetamol tablets
  Interventions: Drug: Paracetamol tablets

INTERVENTIONS:
Drug: Paracetamol hot drink — Hot drink containing paracetamol
  Arms: Paracetamol hot drink
Drug: Paracetamol tablets — Paracetamol tablets
  Arms: Paracetamol tablets

SUMMARY:
The aim of this study is to subjectively assess symptoms in subjects suffering from the common cold following a single dose of paracetamol hot drink compared to paracetamol tablet

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of the common cold of no more than 120 hours duration
* Self-rating congestion of at least moderate severity
* Suffering from at least four symptoms of common cold or flu

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Common Cold Centre, Cardiff, Wales, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: A total of 200 participants were screened and all were randomized into the study.
Groups:
- Mentholated Paracetamol Hot Drink: Mentholated paracetamol hot drink prepared by dissolving 500 milligram (mg) of paracetamol in 200 milliliter (mL) of boiled mineral water was taken orally by participants within a time period of 15 minutes.
- Paracetamol Tablet: Paracetamol 500 mg tablet was taken orally with measured 200 mL of ambient mineral water.
Period: Overall Study
Arm/Group | Mentholated Paracetamol Hot Drink | Paracetamol Tablet
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mentholated Paracetamol Hot Drink: Mentholated paracetamol hot drink prepared by dissolving 500 mg of paracetamol in 200 mL of boiled mineral water was taken orally by participants within a time period of 15 minutes.
- Total: Total of all reporting groups
Arm/Group | Mentholated Paracetamol Hot Drink | Paracetamol Tablet | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.0 (1.85) | 20.0 (1.98) | 20.0 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 63 | 128
  Male | 35 | 37 | 72

OUTCOME MEASURES:

1. Primary Outcome: Breathing Scores Post 15 Minutes
Description: A mean breathing score was calculated at baseline, 30 seconds, 2, 5 and 15 minutes, derived from participant responses to questions relating to breathing i.e. "my breathing feels easy", "I feel airways are open", "I feel a cooling sensation in my throat", "I can feel the air flowing to my lungs easily", "My nose feels less blocked" and "I feel my breathing is comfortable". The breathing scores were rated by the participants on a 5 point (0-4) rating scale with '0' being labeled as 'strongly disagree' and '4' being labeled as 'strongly agree'. For each participant, a mean score was derived by summing the responses and dividing by the number of questions answered.
Time Frame: Baseline to 15 minutes
Population: Intent to Treat (ITT) Population: All randomized participants who had at least one post-baseline efficacy evaluation.
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Mentholated Paracetamol Hot Drink | Paracetamol Tablet
Number analyzed (Participants) | 100 | 100
Score on a Scale | 0.83 [0.73 to 0.93] | 0.11 [0.01 to 0.21]
Statistical Analysis 1: Comparison: Mentholated Paracetamol Hot Drink vs Paracetamol Tablet; Null Hypothesis considered no difference in treatments being compared for breathing score over the first 15 minutes compared to baseline; Test type: Superiority or Other; p < 0.0001, Repeated Measure Analysis; Repeated measures analysis with factors for time and treatment*time interaction. Baseline score was adjusted as part of the repeated measures series; Adjusted Mean difference = 0.72, 95% CI 2-sided [0.58 to 0.86] — Difference was first named treatment minus second named treatment such that a positive difference favours the first named treatment

2. Secondary Outcome: Breathing Score Post 60 Minutes
Description: A mean breathing score was calculated at baseline, 30 seconds, 2, 5, 15 and 60 minutes, derived from participant responses to questions relating to breathing i.e. "my breathing feels easy", "I feel airways are open", "I feel a cooling sensation in my throat", "I can feel the air flowing to my lungs easily", "My nose feels less blocked" and "I feel my breathing is comfortable". The breathing scores were rated by the participants on a 5 point (0-4) rating scale with '0' being labeled as 'strongly disagree' and '4' being labeled as 'strongly agree'. For each participant, a mean score was derived by summing the responses and dividing by the number of questions answered.
Time Frame: Baseline to 60 minutes
Population: ITT population: All randomized participants who had at least one post-baseline efficacy evaluation.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Mentholated Paracetamol Hot Drink | Paracetamol Tablet
Number analyzed (Participants) | 100 | 100
Score on a scale | 0.92 [0.81 to 1.02] | 0.34 [0.23 to 0.44]
Statistical Analysis 1: Comparison: Mentholated Paracetamol Hot Drink vs Paracetamol Tablet; Null hypothesis considered no difference in treatments being compared for breathing score over 60 minutes; Test type: Superiority or Other; p < 0.0001, Repeated measures analysis; [statistical method as in outcome 1, analysis 1]; Adjusted Mean Difference = 0.58, 95% CI 2-sided [0.44 to 0.72] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Cold Symptoms Score Post 15 Minutes
Description: A mean Cold symptom score was calculated at baseline, 30 seconds, 2, 5 and 15 minutes from participant responses to questions relating to cold symptoms i.e. "My head feels clear", "I feel soothing in my throat" and "I feel my cough is being soothed". The cold symptom scores were rated by the participants on a 5 point (0-4) rating scale with '0' being labeled as 'strongly disagree' and '4' being labeled as 'strongly agree'. For each participant, a mean score was derived by summing the responses and dividing by the number of questions answered.
Time Frame: Baseline to 15 minutes
Population: ITT Population: all randomized participants who had at least one post-baseline efficacy evaluation.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Mentholated Paracetamol Hot Drink | Paracetamol Tablet
Number analyzed (Participants) | 100 | 100
Score on a scale | 0.64 [0.52 to 0.75] | 0.13 [0.02 to 0.25]
Statistical Analysis 1: Comparison: Mentholated Paracetamol Hot Drink vs Paracetamol Tablet; Null Hypothesis considered no difference in treatments being compared for cold symptoms score after 60 minutes; Test type: Superiority or Other; p < 0.0001, Repeated measures analysis; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.50, 95% CI 2-sided [0.36 to 0.65] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Cold Symptoms Score Post 60 Minutes
Description: A mean Cold symptom score was calculated at baseline, 30 seconds, 2, 5, 15 and 60 minutes from participant responses to questions relating to cold symptoms i.e. "My head feels clear", "I feel soothing in my throat" and "I feel my cough is being soothed". The cold symptom scores were rated by the participants on a 5 point (0-4) rating scale with '0' being labeled as 'strongly disagree' and '4' being labeled as 'strongly agree'. For each participant, a mean score was derived by summing the responses and dividing by the number of questions answered.
Time Frame: Baseline to 60 minutes
Population: ITT population: all randomized participants who had at least one post-baseline efficacy evaluation.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Mentholated Paracetamol Hot Drink | Paracetamol Tablet
Number analyzed (Participants) | 100 | 100
Score on a scale | 0.87 [0.76 to 0.99] | 0.35 [0.24 to 0.46]
Statistical Analysis 1: Comparison: Mentholated Paracetamol Hot Drink vs Paracetamol Tablet; Null hypothesis considered two treatments being compared to be equal for cold symptom score after 60 minutes; Test type: Superiority or Other; p < 0.0001, Repeated measures analysis; [statistical method as in outcome 1, analysis 1]; Adjusted Mean Difference = 0.52, 95% CI 2-sided [0.38 to 0.67] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Soothing Attribute Scores
Description: Soothing attribute of test treatment was assessed by asking the question "if the hot drink is soothing" at baseline, 15 and 60 minutes. The response to the question was rated by participants on a 5 point (0-4) rating scale with '0' being labeled as 'strongly disagree' and '4' being labeled as 'strongly agree'.
Time Frame: Baseline to 15 and 60 minutes
Population: ITT population: all randomized participants who had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mentholated Paracetamol Hot Drink | Paracetamol Tablet
Number analyzed (Participants) | 100 | 100
Score on a scale
  Average effect over first 15 minutes | 2.3 (0.80) | 1.2 (0.88)
  Average effect over 60 minutes | 2.4 (0.72) | 1.3 (0.88)

6. Secondary Outcome: Overall Cold Symptoms Score
Description: Overall cold symptom score was assessed by asking the question "my cold symptoms are improved" only post consuming the drink at baseline, 15 and 60 minutes . The response to the question was rated by participants on a 5 point (0-4) rating scale with '0' being labeled as 'strongly disagree' and '4' being labeled as 'strongly agree'.
Time Frame: Baseline to 15 and 60 minutes
Population: ITT population: all randomized participants who had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Mentholated Paracetamol Hot Drink | Paracetamol Tablet
Number analyzed (Participants) | 100 | 100
Score on a scale
  Average effect over first 15 minutes | 1.8 (0.86) | 0.9 (0.63)
  Average effect over 60 minutes | 2.1 (0.75) | 1.3 (0.62)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the treatment, and until 5 days following administration of the last dose of investigational product.
Groups:
- Paracetamol Tablets: Paracetamol 500 mg tablet was taken orally with measured 200 mL of ambient mineral water.
Arm/Group | Mentholated Paracetamol Hot Drink | Paracetamol Tablets
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.